CLINICAL TRIAL: NCT03099382
Title: A Randomized, Open-Label, Active-Controlled, Multi-Center, Phase III Clinical Study of Anti-PD-1 Antibody SHR-1210 vs. Investigator's Choice of Chemotherapy in Subjects With Locally Advanced or Metastatic Esophageal Cancer
Brief Title: Study of SHR-1210 Versus Investigator's Choice of Chemotherapy for Participants With Advanced Esophageal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-III-301-ESC
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Results first posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-04

CONDITIONS: Esophageal Carcinoma
MeSH Terms: conditions — Esophageal Neoplasms | interventions — camrelizumab; Docetaxel; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- camrelizumab (Experimental)
  Interventions: Biological: camrelizumab
- Investigator's Choice of Standard Therapy (Active Comparator): Docetaxel or Irinotecan
  Interventions: Drug: Docetaxel; Drug: Irinotecan

INTERVENTIONS:
Biological: camrelizumab — Subjects receive camrelizumab intravenous infusion at the dose 200mg on Day 1 every 2 weeks
  Other Names: SHR-1210
  Arms: camrelizumab
Drug: Docetaxel — Subjects receive Docetaxel intravenous infusion at the dose 75mg/m2 on Day 1 every 3 weeks
  Arms: Investigator's Choice of Standard Therapy
Drug: Irinotecan — Subjects receive Irinotecan intravenous infusion at the dose 180mg/m2 on Day 1 every 2 weeks
  Arms: Investigator's Choice of Standard Therapy

SUMMARY:
In this study, participants with advanced or metastatic squamous cell carcinoma of the esophagus that has progressed after first-line standard therapy will be randomized to receive either single agent SHR-1210 or the Investigator's choice of standard therapy with docetaxel or irinotecan. The primary study hypothesis is that treatment with SHR-1210 will prolong overall survival (OS) as compared to treatment with standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. age: 18-75 years, male or female.
2. Histologically or cytologically confirmed Squamous Cell Carcinoma of the Esophagus, locally advanced, unresectable disease, recurrent or Metastatic disease.
3. Fail to the first-line standard therapy.
4. Measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
5. Can provide either a newly obtained or archival tumor tissue sample.
6. ECOG 0-1.
7. Life expectancy of greater than 12 weeks.
8. Adequate organ function.
9. Female: child bearing potential, a negative urine or serum pregnancy test result within 72 h before study treatment. Participants of reproductive potential must be willing to use adequate contraception for the course of the study through 3 months after the last dose of SHR-1210 or through 180 days after the last dose of docetaxel or irinotecan.
10. Patient has given written informed consent.

Exclusion Criteria:

1. Has a known additional malignancy within the last 5 years before study treatment with the exception of curatively treated basal cell and squamous cell carcinoma of the skin and/or curatively resected in-situ cervical and/or breast cancers.
2. Known central nervous system (CNS) metastases.
3. Subjects with any active autoimmune disease or history of autoimmune disease.
4. Uncontrolled clinically significant heart disease, including but not limited to the following: (1) > NYHA II congestive heart failure; (2) unstable angina, (3) myocardial infarction within the past 1 year; (4) clinically significant supraventricular arrhythmia or ventricular arrhythmia requirement for treatment or intervention;
5. Active infection or an unexplained fever > 38.5°C before two weeks of randomization (subjects with tumor fever may be enrolled at the discretion of the investigator);
6. History of Interstitial Pneumonia or received Corticosteroids for non-infectious pneumonitis.
7. Known Human Immunodeficiency Virus (HIV) infection, active Hepatitis B or Hepatitis C.
8. BMI, <18.5mg/m2 or ≥10% weight lost before screening.
9. Prior therapy with a PD-1, anti-PD-Ligand 1 (PD-L1) agent.
10. Known history of hypersensitivity to macromolecular protein preparation or any components of the SHR-1210 formulation, allergy, hypersensitivity, or contraindication to docetaxel, or irinotecan.
11. Concurrent medical condition requiring the use of cortisol ( >10mg/day Prednisone or equivalent dose) or other systematic immunosuppressive medications within 14 days before the study treatment. Except: inhalation or topical corticosteroids. Doses > 10 mg/day prednisone or equivalent for replacement therapy.
12. Has received prior anti-cancer monoclonal antibody (mAb), chemotherapy, targeted small molecule therapy, or radiation therapy within 4 weeks prior to study Day 1 or not recovered from adverse events due to a previously administered agent.
13. Currently participating or has participated in a study within 4 weeks of the first dose of study medication.
14. Received a live vaccine within 4 weeks of the first dose of study medication.
15. Pregnancy or breast feeding.
16. According to the investigator, other conditions that may lead to stop the research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - 307 Hospital of PLA, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huang J, Xu J, Chen Y, Zhuang W, Zhang Y, Chen Z, Chen J, Zhang H, Niu Z, Fan Q, Lin L, Gu K, Liu Y, Ba Y, Miao Z, Jiang X, Zeng M, Chen J, Fu Z, Gan L, Wang J, Zhan X, Liu T, Li Z, Shen L, Shu Y, Zhang T, Yang Q, Zou J; ESCORT Study Group. Camrelizumab versus investigator's choice of chemotherapy as second-line therapy for advanced or metastatic oesophageal squamous cell carcinoma (ESCORT): a multicentre, randomised, open-label, phase 3 study. Lancet Oncol. 2020 Jun;21(6):832-842. doi: 10.1016/S1470-2045(20)30110-8. Epub 2020 May 13. PMID 32416073

RESULTS

PARTICIPANT FLOW:
Groups:
- Camrelizumab: camrelizumab: Subjects received camrelizumab intravenous infusion at the dose 200mg on Day 1 every 2 weeks
- Investigator's Choice of Standard Therapy: Docetaxel or Irinotecan
  Docetaxel: Subjects received Docetaxel intravenous infusion at the dose 75mg/m2 on Day 1 every 3 weeks
  Irinotecan: Subjects received Irinotecan intravenous infusion at the dose 180mg/m2 on Day 1 every 2 weeks
Period: Overall Study
Arm/Group | Camrelizumab | Investigator's Choice of Standard Therapy
Started | 228 | 220
Completed | 226 | 217
Not Completed | 2 | 3
Not completed — Protocol Violation | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Camrelizumab | Investigator's Choice of Standard Therapy | Total
Number analyzed (Participants) | 228 | 220 | 448
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (7.46) | 59.5 (6.68) | 59.4 (7.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 28 | 48
  Male | 208 | 192 | 400
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 228 | 220 | 448
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 228 | 220 | 448

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Time Frame: approximately 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Camrelizumab | Investigator's Choice of Standard Therapy
Number analyzed (Participants) | 228 | 220
months | 8.28 [6.77 to 9.72] | 6.24 [5.68 to 6.93]

ADVERSE EVENTS:
Time Frame: approximately 24 months
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Camrelizumab | Investigator's Choice of Standard Therapy
All-Cause Mortality (participants affected / at risk) | 23/228 | 10/220
Serious Adverse Events (participants affected / at risk) | 71/228 | 52/220
Other Adverse Events (participants affected / at risk) | 226/228 | 210/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Camrelizumab (N=228) | Investigator's Choice of Standard Therapy (N=220)
Dysphagia (Gastrointestinal disorders) | 4 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 3
Reactive Oral Capillary Endothelial Proliferation (Gastrointestinal disorders) | 2 | 0
Esophageal Obstruction (Gastrointestinal disorders) | 2 | 0
Oesophageal Fistula (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 3
Subileus (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Oesophageal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Pain (Gastrointestinal disorders) | 1 | 0
Gastric Obstruction (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Diaphragmatic Hernia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 5
Nausea (Gastrointestinal disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 1
Noninfective Gingivitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Perforation (Gastrointestinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Oesophagobronchial Fistula (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Tracheal Stenosis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tracheal Mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung Infection (Infections and infestations) | 7 | 7
H1N1 Influenza (Infections and infestations) | 1 | 0
Viral Infection (Infections and infestations) | 1 | 0
Soft Tissue Infection (Infections and infestations) | 1 | 0
Carbuncle (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2
Anal Infection (Infections and infestations) | 0 | 1
Death (General disorders) | 5 | 3
Pyrexia (General disorders) | 3 | 0
Asthenia (General disorders) | 2 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 2 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 4 | 1
Chronic Cholecystitis (Hepatobiliary disorders) | 0 | 1
Reactive Cutaneous Capillary Endothelial Proliferation (Skin and subcutaneous tissue disorders) | 4 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0
Blood Bilirubin Increased (Investigations) | 1 | 0
Blood Calcium Increased (Investigations) | 1 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 6
Neutrophil Count Decreased (Investigations) | 0 | 3
Platelet Count Decreased (Investigations) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Bone Marrow Toxicity (Blood and lymphatic system disorders) | 0 | 2
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 2
Nasal Mucosa Reactive Capillary Endothelial Proliferation (Vascular disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Venous Thrombosis Limb (Vascular disorders) | 0 | 1
Circulatory Collapse (Vascular disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Adrenal Insufficiency (Endocrine disorders) | 1 | 0
Myasthenia Gravis (Nervous system disorders) | 1 | 0
Loss of Consciousness (Nervous system disorders) | 0 | 1
Device Loosening (Product Issues) | 1 | 0
Completed Suicide (Psychiatric disorders) | 1 | 0
Anastomotic Ulcer (Injury, poisoning and procedural complications) | 0 | 1
Drug Hypersensitivity (Immune system disorders) | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Camrelizumab (N=228) | Investigator's Choice of Standard Therapy (N=220)
Anaemia (Blood and lymphatic system disorders) | 102 | 107
Sinus tachycardia (Cardiac disorders) | 13 | 6
Hypothyroidism (Endocrine disorders) | 40 | 11
Hyperthyroidism (Endocrine disorders) | 14 | 2
Constipation (Gastrointestinal disorders) | 39 | 26
Diarrhoea (Gastrointestinal disorders) | 31 | 78
Nausea (Gastrointestinal disorders) | 19 | 87
Vomiting (Gastrointestinal disorders) | 19 | 64
Abdominal distension (Gastrointestinal disorders) | 13 | 9
Abdominal pain upper (Gastrointestinal disorders) | 13 | 6
Oesophageal obstruction (Gastrointestinal disorders) | 12 | 2
Dysphagia (Gastrointestinal disorders) | 11 | 12
Abdominal pain (Gastrointestinal disorders) | 4 | 17
Asthenia (General disorders) | 54 | 75
Pyrexia (General disorders) | 38 | 21
Chest pain (General disorders) | 23 | 19
Oedema peripheral (General disorders) | 12 | 2
Chest discomfort (General disorders) | 9 | 13
Hepatic function abnormal (Hepatobiliary disorders) | 14 | 5
Upper respiratory tract infection (Infections and infestations) | 15 | 11
Weight decreased (Investigations) | 44 | 41
Aspartate aminotransferase increased (Investigations) | 33 | 17
White blood cell count decreased (Investigations) | 33 | 112
Alanine aminotransferase increased (Investigations) | 24 | 18
Bilirubin conjugated increased (Investigations) | 19 | 9
Neutrophil count decreased (Investigations) | 17 | 75
White blood cell count increased (Investigations) | 16 | 4
Neutrophil count increased (Investigations) | 15 | 5
Lymphocyte count decreased (Investigations) | 14 | 10
Platelet count decreased (Investigations) | 14 | 13
Blood bilirubin increased (Investigations) | 12 | 9
Blood albumin decreased (Investigations) | 11 | 15
Haemoglobin decreased (Investigations) | 7 | 16
Hyponatraemia (Metabolism and nutrition disorders) | 49 | 20
Decreased appetite (Metabolism and nutrition disorders) | 44 | 80
Hypoalbuminaemia (Metabolism and nutrition disorders) | 43 | 26
Hypoproteinaemia (Metabolism and nutrition disorders) | 28 | 17
Hypokalaemia (Metabolism and nutrition disorders) | 21 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 18
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 14
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 20 | 9
Insomnia (Psychiatric disorders) | 16 | 7
Proteinuria (Renal and urinary disorders) | 31 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 52 | 31
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 16
Productive cough (Respiratory, thoracic and mediastinal disorders) | 17 | 13
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 15 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 12 | 2
Reactive cutaneous capillary endothelial proliferation (Skin and subcutaneous tissue disorders) | 181 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All clinical study findings and documents will be regarded as confidential. The investigator and members of his/her research team must not disclose such information without prior written approval from the sponsor.

DOCUMENTS (2):
  • Study Protocol (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/82/NCT03099382/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/82/NCT03099382/SAP_001.pdf